CLINICAL TRIAL: NCT01143285
Title: Chimiodiet Study:Impact of Early and Active Nutritional and Dietary Management on grade3 or More Toxicities Induced by Chemotherapy and Targeted Therapies Administered to Patients as First Intention for Non Surgical Metastatic Colorectal Cancer.
Brief Title: Impact of Early and Active Nutritional and Dietary Management grade3 or More Toxicities Induced by Chemotherapy and Targeted Therapies Administered to Patients as First Intention for Non Surgical Metastatic Colorectal Cancer
Acronym: CHIMIODIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: UNICANCER (Other); Centre Leon Berard (Other); Centre Val d'Aurelle (Unknown); University Hospital, Montpellier (Other); Assistance Publique Hopitaux De Marseille (Other); Centre hospitalier de Perpignan (Other); Institut Sainte Catherine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-APN-03
Record Dates: First submitted 2009-07-21; First posted 2010-06-14 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Active nutritional and dietary management; Metastatic colorectal cancer; Non surgical metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I - Early and active nutritional support. (Experimental): During the initial consultation, the dietician will answer the questions of the patient and their family. Patients will be seen regularly in follow-up for weight measurement, serum albumin assay, a 1 or 3 day food record and an evaluation of appetite level. Nutritional counselling is then adjusted accordingly and:Balanced meals are continued if weight is stable and appetite is undiminished.Protein and energy fortification is recommended if weight loss is observed or if food intake decreases between 2 consultations leading to total food intake of less than 50% of required food intake. When a patient presents with signs of malnutrition according to the criteria set out by the Authority for Health, oral nutritional support (ONS) is set up, in agreement with the department head. Two 200ml bottles of Fortimel Extra are to be taken every day. If this ONS strategy is insufficient to improve the patient's nutritional status, artificial nutrition should be discussed.
  Interventions: Other: Early and active nutritional support.
- II - No nutritional support (No Intervention): Should malnutrition develop in a group II patient, ONS will be ordered. It will consist of two 200ml Fortimel Extra* bottles per day in addition to regular meals. Ideally, the ONS should be taken as a snack outside of meal times so as to not spoil the appetite. If this ONS is insufficient to improve the nutritional status of the patient, artificial nutrition (either enteral or parenteral) will be discussed.

INTERVENTIONS:
Other: Early and active nutritional support. — The first nutritional consultation coincides with the 1st CT consultation. An overview of the nutritional support strategy is given, along with specific goals and the twice monthly follow-up schedule that accompanies the chemotherapy courses. The nutritionist once again goes over the various side effects of the medication. Special attention will be given to digestive side effects and their consequences on appetite levels and weight loss during treatment.A qualitative and quantitative 3-day food record will precede the 1st course of CT. This food record is given to patients during the 1st selection visit, in order to evaluate spontaneous oral food intake and dietary habits. Information from the different food groups serves as a starting point for the dietician to explain how to adapt food intake through fortification, portion control according to appetite fluctuations and the onset of side effects.
  Arms: I - Early and active nutritional support.

SUMMARY:
Description of active nutritional support: Early and active nutritional support is mainly concerned with maintaining protein and energy intake levels despite chemotherapy. A part-time nutritionist will be assigned to each research centre. She will cover active nutritional support during a one-hour consultation and assist the investigating oncologist in filling out the e-CRF data. A two-day meeting prior to the beginning of the study will enable the standardization of active nutritional support strategy across all research centres:

* The nutritionist will explain the consequences of the side effects of chemotherapy on appetite levels and nutritional status.
* Spontaneous oral intake and eating habits will be assessed based on a qualitative and quantitative 3-day food record.
* Then the nutritionist will explain to patients how to adapt their diet (fortification, portion control etc.) according to personal preferences and dietary habits, appetite fluctuation and side effects.
* A booklet containing an overview of the nutritional counsel, recipe ideas, an example of a daily menu, energy equivalence tables and specific diet and hygiene tips for each possible side effects of chemotherapy will be given to all patients.
* During each consultation, patients will be weighed, appetite and food intake will be evaluated (24-hour record except for prospective 3-day record of V0, V3, V6, V9, V12, V13 and V14 consultations), chemotherapy side effects will be recorded and nutritional counsel will be adapted to each patient's individual situation. In case of decrease in food intake and/or weight loss, a protein- and energy-rich oral supplement will be given.

In both groups, if a patient exhibits signs of malnutrition (weight loss >5% over a one-month period or > 10% in total) and/or food intake less than 50% of estimated daily requirements, an oral supplement will be given after approval of the oncologist. If this measure is insufficient, artificial nutrition (enteral or parenteral) will be considered.

DETAILED DESCRIPTION:
The "Nutricancer study" carried out on 2,000 French patients showed a malnutrition prevalence rate of 39% in cancer patients. Malnutrition is an independent risk factor for hospital-acquired infections. It also increases the complication rate following surgery, chemotherapy and radiotherapy. It may require a reduction in chemotherapy dosage, thus decreasing the effectiveness of treatment. It increases the length of hospital stays and the cost of care, and has a negative impact on the quality of life of patients (2, 3). Nutritional management is not sufficient. Close to 60% of patients included in the Nutricancer study reported that they had received no nutritional support. Yet, the benefits of nutritional support in perioperative care for surgical colorectal cancers is well established. A recent study suggests that early and active nutritional support in rectal cancer patients reduces the risk of malnutrition, complications from radiotherapy and increases the quality of life of patients. Close to half of patients receiving FOLFOX or FOLFIRI type chemotherapies for metastatic colorectal cancer (CRC) develop a grade 3 toxicity. Our hypothesis is that active nutritional support during chemotherapy for metastatic colorectal cancer will permit the sustainability of intakes and the nutritional status of patients and lead to a reduction in complications, an improvement in quality of life and a reduction in the length of hospital stays.

The goal of our study is to show that early and active nutritional and dietary management (early nutritional support for short) during chemotherapy for metastatic colorectal cancer decreases the risk of malnutrition, reduces chemotherapy toxicity, improves quality of life and decreases the length of hospital stays.

The main evaluation criteria of the study will be the frequency of grade 3 or more toxicity in patients receiving active nutritional support during first line chemotherapy and/or targeted therapy for non surgical metastatic colorectal cancer.

Experimental framework: This is a prospective, multicentre, open, sample-based clinical trial. Patients eligible for the study must have been diagnosed with non surgical metastatic colorectal cancer and be planned to receive 5FU/oxaliplatine or 5FU/irinotecan based chemotherapy, associated or not with targeted therapy. The main exclusion criteria are severe malnutrition, adjuvant radiotherapy, artificial nutrition, pregnancy and breastfeeding, another severe active disease and participation in another clinical trial.

The ChimioDiet study will be proposed during the consultation meant to set up chemotherapy. Selected patients will be randomly assigned to two groups:

* Group I: patients receiving active nutritional support from the first chemotherapy session.
* Group II: patients initially receiving no active nutritional support. Random assignment of patients to groups will be automatically generated by the e-CRF software, taking into account the need for stratification according to research centre and chemotherapy type.

An evaluation of nutritional status will be carried out every two weeks (weight, appetite and intake record). Patients with malnutrition or dietary intakes below 50% of recommended daily intake over 2 consecutive consultations will receive a protein- and calorie-rich oral supplement or, if required, enteral or parenteral artificial nutrition. All undesirable effects of chemotherapy will be recorded. Patients will be required to fill out a quality of life questionnaire (EORTC QLQ-C30) upon selection for inclusion in the study and every three months thereafter.

The analysis of the main judgement criteria will rely on a logistic regression. Measured outcome will be the occurrence of a grade 3 or more toxicity. The main explanatory variables will be the group to which the patient has been assigned (early and active nutritional support or not). The analysis will also take into account the main stratification parameters, namely treatment centre and type of chemotherapy.

Description of active nutritional support: Early and active nutritional support is mainly concerned with maintaining protein and energy intake levels despite chemotherapy. A part-time nutritionist will be assigned to each research centre. She will cover active nutritional support during a one-hour consultation and assist the investigating oncologist in filling out the e-CRF data. A two-day meeting prior to the beginning of the study will enable the standardization of active nutritional support strategy across all research centres:

* The nutritionist will explain the consequences of the side effects of chemotherapy on appetite levels and nutritional status.
* Spontaneous oral intake and eating habits will be assessed based on a qualitative and quantitative 3-day food record.
* Then the nutritionist will explain to patients how to adapt their diet (fortification, portion control etc.) according to personal preferences and dietary habits, appetite fluctuation and side effects.
* A booklet containing an overview of the nutritional counsel, recipe ideas, an example of a daily menu, energy equivalence tables and specific diet and hygiene tips for each possible side effects of chemotherapy will be given to all patients.
* During each consultation, patients will be weighed, appetite and food intake will be evaluated (24-hour record except for prospective 3-day record of V0, V3, V6, V9, V12, V13 and V14 consultations), chemotherapy side effects will be recorded and nutritional counsel will be adapted to each patient's individual situation. In case of decrease in food intake and/or weight loss, a protein- and energy-rich oral supplement will be given.

In both groups, if a patient exhibits signs of malnutrition (weight loss >5% over a one-month period or > 10% in total) and/or food intake less than 50% of estimated daily requirements, an oral supplement will be given after approval of the oncologist. If this measure is insufficient, artificial nutrition (enteral or parenteral) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients with synchrone or metachronous CRC metastases without possible initial surgical outcome
* Patients covered by Social Security
* Patients willing to sign the proper consent forms

Exclusion Criteria:

* Severely malnourished patients according to the Authority for Health criteria : weight loss > 5% of base weight in less than one month or > 10% of base weight in less than six months and/or BMI < 18 or 21.5 in patients 70 years old or more, and/or serum albumin assay < 35 g/l.
* Patients receiving concomitant radiotherapy.
* Patients receiving or programmed to receive artificial nutrition (enteral or parenteral).
* Pregnant or breastfeeding women (a qualitative urine pregnancy test will be given to all women of child-bearing age).
* Patients incapable of understanding (foreign language, intellectual deficiencies, motor cortex deficiencies...) and/or applying the nutritional counselling (persons institutionalised in a rest home, retirement home, prison etc.).
* Patients with another sever debilitating disease likely to impact on nutritional status (cardiac, hepatic, or renal insufficiency etc.).
* Persons already participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Toxicities frequently associated with chemotherapy | 2 weeks
  Number and grade of: diarrhoea,nausea,vomiting, oral mucositis,fatigue, neurotoxicities, dysgeusia,haematological toxicities such as leukopenia neutropenia,anemia and thrombocytopenia.

SECONDARY OUTCOMES:
Nutritional status of patients | 2 weeks
  Measures: weight, body mass index
Appetite measures | 2 weeks
  Spontaneous food intake, EVA
Quality of life | 3 months
  questionary EORTC QLQ-C30
Number of occurrences of grades 1 and 2 toxicities | 2 weeks
The number of hospital days | All study
Overall survival | All study

CONTACTS AND LOCATIONS:
Overall Officials: Xavier HEBUTERNE, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (8):
- France (8):
  - Institut Sainte Catherine, Avignon
  - The Léon Bérard Cancer Centre, Lyon
  - Assistance Publique des hopitaux de Marseille, Marseille
  - The Val d'Aurelle Cancer Centre, Montpellier
  - University Hospital, Montpellier, Montpellier
  - The Antoine Lacassagne Cancer Centre, Nice
  - The digestive oncology departement of the Archet Hospital of the Nice University Hospital Centre, Nice
  - Hospital in Perpignan, Perpignan

REFERENCES:
- [Background] 1. Situation du cancer en France en 2007 - Synthèses rapports INCa - http://www.e-cancer.fr 2.Dewys et al.,Pronostic effect of weight loss prior to CT in cancer patient. Am J.Med 1980; 69 (4): 491-7; 3. Étude Nutricancer 2005, Hébuterne et al, Nutr Clin Metabol 2006.4.Gupta D, Lis CG, Granick J, Grutsch JF, Vashi PG, Lammersfeld CA. Malnutrition associated with poor quality of life in CR cancer:retrospective analysis.J Clin Epidemiol 2006 Jul;59(7):704-9. Epub 2006 Apr 19. 5. Andreyev et al., Why do patients with weight loss have a worse outcome when undergoing CT for gastrointestinal malignancies, Eur J Cancer 1998 Mar; 34(4): 503-9;6. Schneider et al, Malnutrition is an independant factor associated with nosocomial infections, Br J Nutr 2004 Jul; 92(1): 105-11. 7.Tucker HN, Miquel SG. : cost containment through nutrition intervention. Nutr Rev 1996 Apr; 54: 111-21.8. Colucci G, Gebbia V, Paoletti G, Giuliani F, Caruso M, Gebbia N et al . Gruppo Oncologico Dell'Italia Meridionale. Phase III randomized trial of FOLFIRI VS FOLFOX4 in the treatment of advanced CCR: a multicenter study of the Gruppo Oncologico Dell'Italia Meridionale. J Clin Oncol. 2005 Aug 1;23(22):4866-75. Epub 2005 Jun 6.9. Douillard JY, Sobrero A, Carnaghi C, Comella P, Díaz-Rubio E, Santoro A et al. Metastatic CR cancer: integrating irinotecan into combination and sequential CT. Ann Oncol. 2003;14 Suppl 2:ii7-12. Review.10. Hurwitz HI, Fehrenbacher L, Hainsworth JD, Heim W, Berlin J, Holmgren E et al. Bevacizumab in combination with fluorouracil and leucovorin: an active regimen for first-line metastatic colorectal cancer.J Clin Oncol. 2005 May 20;23(15):3502-8.11. Saltz LB, Meropol NJ, Loehrer PJ Sr, Needle MN, Kopit J, Mayer RJ. Phase II trial of cetuximab in patients with refractory CR cancer that expresses the epidermal growth factor receptor. J Clin Oncol. 2004 Apr 1;22(7):1201-8. Epub 2004 Mar 1
- See also: Situation du cancer en France en 2007 - Synthèses rapports INCa — http://www.e-cancer.fr